CLINICAL TRIAL: NCT00709618
Title: A Phase II, Single-Arm, Multi-Center Study Evaluating the Combination of Vinorelbine and Lapatinib in Women With ErbB2 Overexpressing Metastatic Breast Cancer
Brief Title: Lapatinib + Vinorelbine in ErbB2 Overexpressing, First or Second Line Metastatic Breast Cancer Subjects
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Evolving standard of care practices in this disease setting was limiting enrolment and leading to a delay in delivering this study information to the public.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LPT111110
Record Dates: First submitted 2008-07-02; First posted 2008-07-03 (Estimated); Results first posted 2013-01-18 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-06

CONDITIONS: Neoplasms, Breast
Keywords: Erbb2; MBC; First or Second line therapy; Metastatic Breast Cancer; Vinorelbine; Tykerb
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Lapatinib, Vinorelbine — Vinorelbine intravenously once weekly for 3 weeks, followed by a rest week in a 4-week cycle) plus lapatinib daily
  Other Names: Lapatinib; Vinorelbine

SUMMARY:
This is an open-label, single-arm, multi-center, Phase II study to determine the activity of vinorelbine plus lapatinib in either first- or second-line setting in women with ErbB2 overexpressing metastatic breast cancer (MBC). Sixty subjects will be enrolled in the study. Subjects will receive vinorelbine intravenously once weekly for 3 weeks, followed by a rest week in a 4-week cycle) plus lapatinib daily. Subjects will receive treatment until disease progression or withdrawal from the study. The primary objective of this study is to evaluate overall tumor response rate of lapatinib in combination with vinorelbine. Secondary objectives include progression-free survival, overall survival, duration of response, time to response and time to progression and safety. Safety and efficacy assessments will be performed at 4, 8 and 12 week intervals, and at the end of treatment.

Subject: Metastatic Breast Cancer, ErbB2, First-line or Second-line therapy, Lapatinib, Vinorelbine

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for inclusion in this study only if all of the following criteria apply:

1. Signed informed consent prior to registration.
2. Considered by the Investigator to have a life expectancy of ≥12 weeks.
3. Subjects must have histologically confirmed invasive breast cancer with Stage IV disease at primary diagnosis or at relapse after curative-intent surgery.

   • Where the disease is restricted to a solitary lesion, the neoplastic nature of the lesion should be confirmed by cytology or histology.
4. Documented amplification of ErbB2 3+ by immunohistochemistry or a positive score (>2.2) by fluorescence in situ hybridization (FISH) using a local laboratory result (which will be considered sufficient in this study with no further verification by a central laboratory). NOTE: If both IHC and FISH results available, FISH results must be used for eligibility.
5. Subjects must not have received more than 1 prior chemotherapeutic regimen in the metastatic setting.
6. All prior chemotherapy, immunotherapy, biologic therapy, or surgery (except for minor surgical procedures) must be discontinued at least 4 weeks prior to first dose of investigational product. Hormonal therapy must be discontinued at least 1 week prior to first dose.
7. Prior diagnosis of cancer is allowed as long as the subject is free of disease and has been off treatment for prior malignancies for 5 years. Subjects with completely resected basal or squamous cell skin cancer or successfully treated cervical carcinoma in situ will be allowed if it has been 1 year or longer since definitive surgery.
8. Subjects must have measurable disease, according to Response Evaluation Criteria in Solid Tumors (RECIST) guidelines.
9. Females aged ≥18 years with any menopausal status:

   * Non-child-bearing potential (i.e., women with functioning ovaries who have a current documented tubal ligation or hysterectomy, or women who are postmenopausal)
   * Child-bearing potential (i.e., women with functioning ovaries and no documented impairment of oviductal or uterine function that would cause sterility): This category includes women with oligomenorrhea (severe), women who are perimenopausal, and young women who have begun to menstruate. These subjects must have a negative serum pregnancy test at screening and agree to one of the following:
   * Complete abstinence from intercourse from 2 weeks prior to administration of the first dose of study medication until 28 days after the final dose of study medication; or
   * Consistent and correct use of one of the following acceptable methods of birth control: male partner who is sterile prior to the female subject's entry into the study and is the sole sexual partner for that female subject; any intrauterine device with a documented failure rate of less than 1% per year; oral contraceptives (either combined or progestogen only) where not contraindicated for this subject population or per local practice.; or barrier methods, including diaphragm or condom with a spermicide.
10. ECOG performance status (PS) of 0 to 2 [Oken, 1982] (Appendix 1).
11. Subjects must have normal organ and marrow function as defined in Table 1. Table 1 Baseline Laboratory Values for Adequate Organ Function System Laboratory Value Hematologic Absolute neutrophil count ≥1.5 × 10^9/L Hemoglobin ≥9 g/dL Platelets ≥100 × 10^9/L Hepatic Serum bilirubin ≤1.25 × upper limit of normal (ULN) Aspartate aminotransferase and alanine aminotransferase

    * 3 × ULN without liver metastases
    * 5 × ULN if documented liver metastases Renal Serum creatinine ≤1.5 mg/dL

      * OR - Calculated creatinine clearance ≥40 mL/min
12. Subjects must have a cardiac ejection fraction of at least 50% (as measured by echocardiogram [ECHO] or multigated acquisition scan [MUGA]) and within the institutional range of normal. Subjects who require cardiac medications (e.g. positive inotropic agents or afterload reducers) for abnormal ejection fraction are ineligible. MUGA scans will be accepted in cases where an ECHO cannot be performed or is inconclusive. The same modality to assess cardiac ejection fraction must be used consistently throughout the study.
13. Radiotherapy prior to initiation of study medication is allowed to a limited area (e.g., palliative therapy), if it is not the sole site of disease. Subjects must have completed radiation treatment and recovered from all acute radiation treatment-related toxicities (e.g., bone marrow suppression) prior to commencement of combination treatment.
14. Subjects with stable central nervous system (CNS) metastases. Subjects with stable CNS metastases are defined as follows: subject is asymptomatic with CNS metastases that have been stable for at least 3 months as confirmed by computed tomography (CT)/magnetic resonance imaging (MRI). Subjects with evidence of leptomeningeal/parenchymal involvement are eligible only if they are not taking steroids or enzyme-inducing anticonvulsants within 4 weeks of commencement of the study. Treatment with prophylactic anticonvulsants is permitted, unless listed as a prohibited medication.
15. Subject must be free of gastrointestinal diseases that impede swallowing and retaining of oral medications.
16. Able to swallow and retain oral medication (intact pill).
17. Bisphosphonate therapy for bone metastases is allowed; however, treatment must be initiated prior to the first dose of study medication. Prophylactic use of bisphosphonates in subjects without bone disease, except for the treatment of osteoporosis, is not permitted.
18. Subjects whose disease is estrogen receptor + and/or progesterone receptor + or unknown status will only be included in the study if they meet the following criteria:

    * They have symptomatic visceral disease that requires chemotherapy.
    * The disease is considered by the Investigator to be progressing rapidly or is life threatening.
    * Subjects who have received endocrine therapy and who are no longer benefiting from this therapy.

Exclusion Criteria:

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

1. Subjects taking treatment with medications provided in the list of restricted medications and substances in the drug information section for lapatinib are not eligible for the study. This includes human immunodeficiency virus-positive subjects receiving combination anti-retroviral therapy because of possible pharmacokinetic interactions with lapatinib.
2. Prior therapy with lapatinib.
3. Prior therapy with vinorelbine for treatment of breast cancer.
4. More than 1 line of therapy for treatment of MBC.
5. Concurrent anticancer or concomitant radiotherapy treatment.
6. History of uncontrolled or symptomatic angina; history of arrhythmias requiring medications; clinically significant myocardial infarction <6 months from study entry; uncontrolled or symptomatic congestive heart failure; ejection fraction below the institutional normal limit; or any other cardiac condition, which in the opinion of the treating physician, would make this protocol unreasonably hazardous for the patient.
7. Have current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment)
8. Use of an investigational drug within 30 days or 5 half-lives, whichever is longer, preceding the first dose of investigational treatment, or, concurrent treatment with an investigational agent or participation in another clinical trial involving investigational agents.
9. Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to any of the agents used in this study or their excipients.
10. Known history of uncontrolled inter-current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, clinically significant cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
11. Concurrent disease or condition that would make the woman inappropriate for study participation, or any serious medical disorder that would interfere with the woman's safety.
12. Pregnant or lactating females at any time during the study (due to the potential teratogenic or abortifacient effects of lapatinib and breastfeeding).
13. Subjects with diseases affecting gastrointestinal function resulting in an inability to take oral medication, including; malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel.

    Women with ulcerative colitis are also excluded.
14. Peripheral neuropathy of Grade 2 or greater.
15. Unresolved or unstable, serious toxicity from prior administration of another investigational drug and/or of prior cancer treatment.
16. Dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2008-06; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (22):
- United States (22):
  - GSK Investigational Site, Muscle Shoals, Alabama
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Plantation, Florida
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Cedar Rapids, Iowa
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Bethesda, Maryland
  - GSK Investigational Site, Jackson, Mississippi
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Eugene, Oregon
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Memphis, Tennessee

RESULTS

PARTICIPANT FLOW:
Groups:
- Vinorelbine 20 mg/m^2 Plus Lapatinib 1500 mg: Participants received vinorelbine (20 milligrams per meters squared [mg/m^2]) intravenously (IV) once weekly for 3 weeks (on Days 1, 8, and 15 of a 4-week cycle, followed by a rest week) plus oral lapatinib (1500 mg once daily). Participants received study treatment until disease progression or withdrawal.
Period: Overall Study
Arm/Group | Vinorelbine 20 mg/m^2 Plus Lapatinib 1500 mg
Started | 44
Completed | 14
Not Completed | 30
Not completed — Withdrawal by Subject | 4
Not completed — Lost to Follow-up | 1
Not completed — Study Closed/Terminated | 25

BASELINE CHARACTERISTICS:
Groups:
- Vinorelbine 20 mg/m^2 Plus Lapatinib 1500 mg: Participants received vinorelbine (20 mg/m^2) IV once weekly for 3 weeks (on Days 1, 8, and 15 of a 4-week cycle, followed by a rest week) plus oral lapatinib (1500 mg once daily). Participants received study treatment until disease progression or withdrawal.
Arm/Group | Vinorelbine 20 mg/m^2 Plus Lapatinib 1500 mg
Number analyzed (Participants) | 44
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.2 (12.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 32
  African American/African Heritage | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Overall Response (OR), as Assessed by the Investigator
Description: OR is defined as the number of participants achieving either a confirmed complete response (CR: the disappearance of all target lesions [TLs]) or partial response (PR: a >=30% decrease in the sum of the longest diameter [LD] of the TLs, taking as a reference the baseline sum LD) as assessed by the investigator as the best OR. The best OR is the best response recorded from the start of treatment until disease progression (PD: a >=20% increase in the sum of the LD of TLs, taking as a reference the smallest sum LD recorded since treatment started or the appearance of >=1 new lesions)/recurrence.
Time Frame: From the start of study medication until disease progression, assessed every 8 weeks for up to 2 years
Population: Intent-to-Treat (ITT) Population: participants who received >=1 dose of investigational product. To be assigned a status of PR/CR, a confirmatory disease assessment (including bone scan/positron emission tomography scan documenting that progression/ new lesions hasn't occurred) had to be performed >=4 weeks after response criteria were first met.
Measure: Number; unit: participants
Arm/Group | Vinorelbine 20 mg/m^2 Plus Lapatinib 1500 mg
Number analyzed (Participants) | 44
participants | 18
Statistical Analysis 1: Comparison: Vinorelbine 20 mg/m^2 Plus Lapatinib 1500 mg; Test type: Superiority or Other; percentage of participants = 41, 95% CI 2-sided [26.4 to 55.4] — The estimated value respresents the percentage of participants with a complete response or a partial response

2. Secondary Outcome: Progression-Free Survival (PFS), as Assessed by the Investigator
Description: PFS is defined as the time from the start of treatment until the earliest date of disease progression (PD) or death due to any cause, if sooner. PD is defined as at least a 20% increase in the sum of the LD of target lesions, taking as a reference the smallest sum LD recorded since the treatment started or the appearance of 1 or more new lesions.
Time Frame: From the start of study medication until disease progression, assessed every 8 weeks for up to 2 years
Population: ITT Population. Participants who had neither progressed nor died were censored at the date of the last adequate tumor assessment at the time of the cut-off. Censoring is defined as being alive without the event of interest (progression or death).
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Vinorelbine 20 mg/m^2 Plus Lapatinib 1500 mg
Number analyzed (Participants) | 44
weeks | 24.1 [16.9 to 36.7]

3. Secondary Outcome: Duration of Response, as Assessed by the Investigator
Description: Duration of response, for the subset of participants who had a confirmed CR (the disappearance of all TLs) or PR (a >=30% decrease in the sum of the LD of the TLs, taking as a reference the baseline sum LD), is defined as the time from the first documented evidence of CR or PR until the first documented sign of disease progression (a >=20% increase in the sum of the LD of TLs, taking as a reference the smallest LD recorded since treatment started or the appearance of >=1 new lesions) or death due to any cause, if sooner.
Time Frame: From the start of study medication until disease progression, assessed every 8 weeks for up to 2 years
Population: ITT Population. Only participants with a confirmed CR/PR were assessed for duration of response. To be assigned a status of PR/CR, a confirmatory disease assessment (including bone scan/positron emission tomography scan documenting that progression/ new lesions hasn't occurred) had to be performed >=4 weeks after response criteria were first met.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Vinorelbine 20 mg/m^2 Plus Lapatinib 1500 mg
Number analyzed (Participants) | 18
weeks | 32 [18.0 to 42.3]

4. Secondary Outcome: Time to Response, as Assessed by the Investigator
Description: Time to response, for the subset of participants who had a confirmed CR (the disappearance of all TLs) or PR (a >=30% decrease in the sum of the LD of the TLs, taking as a reference the baseline sum LD), is defined as the time from the start of treatment until the first documented evidence of CR or PR (whichever status was recorded first). When tumor response was confirmed at a repeat assessment, the time to response was taken to be the first time that the response was observed.
Time Frame: From the start of study medication until disease progression, assessed every 8 weeks for up to 2 years
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Vinorelbine 20 mg/m^2 Plus Lapatinib 1500 mg
Number analyzed (Participants) | 18
weeks | 7.5 [7.1 to 8.1]

5. Secondary Outcome: Time to Progression (TTP), as Assessed by the Investigator
Description: TTP is defined as the time from the start of treatment until the earliest date of disease progression (a >=20% increase in the sum of the LD of TLs, taking as a reference the smallest LD recorded since treatment started or the appearance of >=1 new lesions) or death due to breast cancer, if sooner.
Time Frame: From the start of study medication until disease progression, assessed every 8 weeks for up to 2 years
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Vinorelbine 20 mg/m^2 Plus Lapatinib 1500 mg
Number analyzed (Participants) | 44
weeks | 24.1 [16.9 to 36.7]

6. Secondary Outcome: Number of Participants With the Indicated Adverse Events Occurring in at Least 5 Participants and Related to the Combination of Lapatinib and Vinorelbine
Description: Qualitative and quantitative toxicities associated with the combination of lapatinib and vinorelbine during the study are those adverse events (AEs) that are judged to be related to the study treatment by the investigator. Those AEs occuring in more than 5 participants in the ITT Population are listed here.
Time Frame: From the start of study medication until disease progression, assessed every 4 weeks for up to 2 years
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Vinorelbine 20 mg/m^2 Plus Lapatinib 1500 mg
Number analyzed (Participants) | 44
participants
  Diarrhoea | 34
  Nausea | 24
  Constipation | 11
  Vomiting | 9
  Abdominal pain | 7
  Stomatitis | 5
  Neutropenia | 29
  Anaemia | 9
  Fatigue | 20
  Mucosal inflammation | 7
  Rash | 20
  Neutrophil count decreased | 7
  Haemoglobin decreased | 6
  White blood cell count decreased | 5
  Neuropathy peripheral | 5
  Arthralgia | 6
  Decreased appetite | 8

7. Secondary Outcome: Overall Survival
Description: OS is defined as the time from the start of study treatment to the date of death. In the absence of confirmation of death, survival time was to be censored at the last date the participant was known to be alive. Overall survival was not assessed because the study was terminated due to low screening and a low enrollment rate after 3 years. There were no-survival follow-up visits required.
Time Frame: From the start of study treatment to the date of death, assessed for up to 3 years
Arm/Group | Vinorelbine 20 mg/m^2 Plus Lapatinib 1500 mg
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the date of the first dose of study treatment until 30 days post last dose (up to 2 years after the start of the study).
Description: SAEs and non-serious AE data are reported for the ITT Population, comprised of all participants who received at least one dose of investigational product.
Arm/Group | Vinorelbine 20 mg/m^2 Plus Lapatinib 1500 mg
Serious Adverse Events (participants affected / at risk) | 22/44
Other Adverse Events (participants affected / at risk) | 44/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vinorelbine 20 mg/m^2 Plus Lapatinib 1500 mg (N=44)
Neutropenia (Blood and lymphatic system disorders) | 15
Febrile neutropenia (Blood and lymphatic system disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Asthenia (General disorders) | 1
Fatigue (General disorders) | 1
Pyrexia (General disorders) | 1
Perirectal abscess (Infections and infestations) | 1
Viral upper respiratory tract infection (Infections and infestations) | 1
Left ventricular dysfunction (Cardiac disorders) | 1
Blood creatinine increased (Investigations) | 1
Renal failure acute (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vinorelbine 20 mg/m^2 Plus Lapatinib 1500 mg (N=44)
Diarrhoea (Gastrointestinal disorders) | 36
Nausea (Gastrointestinal disorders) | 27
Constipation (Gastrointestinal disorders) | 15
Vomiting (Gastrointestinal disorders) | 14
Abdominal pain (Gastrointestinal disorders) | 10
Dyspepsia (Gastrointestinal disorders) | 8
Stomatitis (Gastrointestinal disorders) | 6
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4
Gastritis (Gastrointestinal disorders) | 3
Mouth ulceration (Gastrointestinal disorders) | 3
Abdominal pain upper (Gastrointestinal disorders) | 2
Abdominal discomfort (Gastrointestinal disorders) | 1
Glossitis (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Lip pain (Gastrointestinal disorders) | 1
Lip swelling (Gastrointestinal disorders) | 1
Oedema mouth (Gastrointestinal disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 1
Proctalgia (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 29
Anaemia (Blood and lymphatic system disorders) | 11
Febrile neutropenia (Blood and lymphatic system disorders) | 3
Leukopenia (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Fatigue (General disorders) | 23
Mucosal inflammation (General disorders) | 7
Pyrexia (General disorders) | 7
Pain (General disorders) | 3
Chest pain (General disorders) | 2
Inflammation (General disorders) | 2
Medical device complication (General disorders) | 2
Non-cardiac chest pain (General disorders) | 2
Oedema peripheral (General disorders) | 2
Application site vesicles (General disorders) | 1
Asthenia (General disorders) | 1
Axillary pain (General disorders) | 1
Catheter site inflammation (General disorders) | 1
Chills (General disorders) | 1
Device infusion issue (General disorders) | 1
Face oedema (General disorders) | 1
Ill-defined disorder (General disorders) | 1
Influenza like illness (General disorders) | 1
Infusion site erythema (General disorders) | 1
Infusion site pain (General disorders) | 1
Local swelling (General disorders) | 1
Malaise (General disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 22
Pruritus (Skin and subcutaneous tissue disorders) | 5
Alopecia (Skin and subcutaneous tissue disorders) | 3
Skin chapped (Skin and subcutaneous tissue disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 2
Nail disorder (Skin and subcutaneous tissue disorders) | 2
Onychoclasis (Skin and subcutaneous tissue disorders) | 2
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2
Night sweats (Skin and subcutaneous tissue disorders) | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Swelling face (Skin and subcutaneous tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4
Pain in jaw (Musculoskeletal and connective tissue disorders) | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1
Urinary tract infection (Infections and infestations) | 6
Upper respiratory tract infection (Infections and infestations) | 5
Sinusitis (Infections and infestations) | 3
Vulvovaginal mycotic infection (Infections and infestations) | 3
Infection (Infections and infestations) | 2
Oral candidiasis (Infections and infestations) | 2
Abscess limb (Infections and infestations) | 1
Acarodermatitis (Infections and infestations) | 1
Breast infection (Infections and infestations) | 1
Candidiasis (Infections and infestations) | 1
Carbuncle (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Fungal skin infection (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 1
Perirectal abscess (Infections and infestations) | 1
Subcutaneous abscess (Infections and infestations) | 1
Viral upper respiratory tract infection (Infections and infestations) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 12
Decreased appetite (Metabolism and nutrition disorders) | 10
Dehydration (Metabolism and nutrition disorders) | 8
Hyponatraemia (Metabolism and nutrition disorders) | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Neutrophil count decreased (Investigations) | 7
Haemoglobin decreased (Investigations) | 6
Weight decreased (Investigations) | 6
White blood cell count decre (Investigations) | 5
Blood creatinine increased (Investigations) | 3
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Blood alkaline phosphatase increased (Investigations) | 2
Lymphocyte count decreased (Investigations) | 2
Blood bilirubin increased (Investigations) | 1
Blood potassium decreased (Investigations) | 1
Blood urea increased (Investigations) | 1
Breath sounds abnormal (Investigations) | 1
White blood cell count increased (Investigations) | 1
Dizziness (Nervous system disorders) | 6
Headache (Nervous system disorders) | 5
Neuropathy peripheral (Nervous system disorders) | 5
Peripheral sensory neuropathy (Nervous system disorders) | 4
Dysgeusia (Nervous system disorders) | 3
Paraesthesia (Nervous system disorders) | 3
Ataxia (Nervous system disorders) | 2
Somnolence (Nervous system disorders) | 2
Burning sensation (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Restless legs syndrome (Nervous system disorders) | 1
Sedation (Nervous system disorders) | 1
Sinus headache (Nervous system disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1
Insomnia (Psychiatric disorders) | 11
Depression (Psychiatric disorders) | 2
Anxiety (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 1
Hallucination (Psychiatric disorders) | 1
Mood altered (Psychiatric disorders) | 1
Restlessness (Psychiatric disorders) | 1
Tearfulness (Psychiatric disorders) | 1
Hot flush (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Jugular vein distension (Vascular disorders) | 1
Lymphoedema (Vascular disorders) | 1
Subclavian vein thrombosis (Vascular disorders) | 1
Diplopia (Eye disorders) | 1
Lacrimation increased (Eye disorders) | 1
Vitreous floaters (Eye disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Ear pain (Ear and labyrinth disorders) | 2
Cholelithiasis (Hepatobiliary disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Seasonal allergy (Immune system disorders) | 2
Left ventricular dysfunction (Cardiac disorders) | 1
Cushingoid (Endocrine disorders) | 1
Thermal burn (Injury, poisoning and procedural complications) | 1
Breast pain (Reproductive system and breast disorders) | 1

LIMITATIONS AND CAVEATS:
The study was terminated due to low screening and a low enrollment rate after 3 years.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.